CLINICAL TRIAL: NCT04424342
Title: Validity and Reliability of the Turkish Version of the Child Perceptions Questionnaire (CPQ8-10)
Brief Title: Turkish Version of the Child Perceptions Questionnaire 8-10
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazife Begüm KARAN, Assistant Professor, DDS, PhD, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 71
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Dentist-Patient Relations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pre-test procedure — The Turkish version of CPQ8-10 was subjected to a preliminary test on a group of 20 children, who were not included in the final study, in order to discuss the intelligibility of the items and to determine comprehension problems for children of this age group
Other: Test re-test — The Turkish version of CPQ8-10 was administered to 50 children who were asked to complete the questionnaire on their own without any assistance. These 50 children were interviewed for a second time within two weeks to measure the reliability of the test-retest

SUMMARY:
The Child Perceptions Questionnaire (CPQ) is a widely used reliable measurement that provides for practitioners to assess child's current emotional, social, and functional well-being. The aim of the present study was to develop a translated version of CPQ8-10 into Turkish language and evaluate its reliability, validity, and reproducibility.

DETAILED DESCRIPTION:
The CPQ8-10 was translated into Turkish as recommended in the literature. The intraclass correlation coefficient (ICC) was used for the test-retest reliability. The internal consistency was evaluated using Cronbach's alpha Coefficient. Construct validity and discriminant validity were calculated, exploratory factor analysis (EFA) and confirmatory factor analysis (CFA) were employed.

ELIGIBILITY:
Inclusion Criteria:

* being aged between 8 and 10 years,
* being mentally and physically sufficient to complete the questionnaire,
* having volunteered to participate in the study,
* speaking Turkish fluently,
* children who were attending their first visit to the dentist

Exclusion Criteria:

* those who were outside this age range (8-10),
* had physical, mental or systemic disabilities that prevented them from understanding and answering the CPQ8-10

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cross-sectional study. Patients applied for RTE University, Department of Pediatric Dentisry
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the penultimate Turkish version of The Child Perceptions Questionnaire 8-10 | 1 day
  The questionnaire has two general questions about the sex and age of the child. The CPQ8-10 was originally composed of 25 items. Responses are recorded using a Likert scale ranging from 1 to 4: "Never"=0; "Once or twice"=1; "Sometimes"=2; "Often"=3; and "Every day or almost every day"=4. The total CPQ8-10 score is calculated by summing all items from four domains, which ranges from 0 to 100, with higher scores indicating worse oral health quality of life and lower scores indicating better oral health quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Nazife Begüm KARAN, Ankara, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Beginning 3 months and ending 5 years following article publication all data can be shared with other researchers